CLINICAL TRIAL: NCT01871233
Title: An Extended Access Program for Perampanel
Status: No longer available | Type: Expanded Access
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E2007-G000-401
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2020-04-16 (Actual); Status verified 2020-03

CONDITIONS: Partial Onset Seizures
Keywords: anti-epileptic drug; Extended Access Program; partial onset seizures; Perampanel
MeSH Terms: interventions — perampanel

INTERVENTIONS:
Drug: Perampanel — Patients will enter this program on the same dose of perampanel that they were receiving at the end of their participation in Studies 207, 307, or 235. Doses of perampanel and of concomitant anti-epileptic drugs (AEDs) can be adjusted based on clinical judgment. A minimum daily dose permitted will be 12 mg per day. Treatment will be prescribed as long as clinically appropriate according to the judgment of the treating physician and the approved summary of Product Characteristics (SmPC). Tablets will be available in strengths of 2 mg, 4 mg, 6 mg, 8 mg, 10 mg, and 12 mg. Patients will be instructed to take their perampanel tablets once daily, by mouth, before bedtime, and with food.
  Other Names: E2007

SUMMARY:
The Extended Access Program (EAP) is a managed access programme for Perampanel. The main objective of this EAP is to ensure that patients participating in studies E2007-A001-207, E2007-G000-307, or E2007-G000-235 continue to have access to perampanel until such time perampanel tablets become commercially available for the treatment of Partial Onset Seizures (POS) in the country in which they reside. This EAP will consist of 2 phases:

* Screening: The patient will start the program once the Screening assessments are completed and the patient is qualified for participation.
* Treatment: Additional assessments, physical examinations, and dosage changes will be clinically determined by the treating physician.

Patients will enter this program on the same dose of perampanel that they were receiving at the end of their participation in previous study. Doses of perampanel and of concomitant anti-epileptic drugs (AEDs) can be adjusted (i.e., added,removed, or changed in dose) based on clinical judgment.

Treatment will be prescribed as long as clinically appropriate according to the judgement of the treating physician and the approved Summary of Product Characteristics (SmPC).

The program will complete in a staggered fashion, country by country, as and when perampanel becomes commercially available for the treatment of POS in each country.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are participating in either Study 207, Study 307, or Study 235 and who in the opinion of the treating physician, continue to benefit from treatment with perampanel (revised per Amendment 01)
* Patients who provide informed consent where applicable per local requirements.
* Female patients of childbearing potential must agree for the duration of the program and for a period of at least 1 month following last dose of perampanel to be abstinent or to commit to the consistent and correct use of a medically acceptable method of birth control (e.g., a double-barrier method [condom plus spermicide, condom plus diaphragm with spermicide])

Exclusion Criteria:

* Patients residing in countries where perampanel is commercially available for the treatment of POS
* Female patients who are lactating, pregnant, or planning to become pregnant

Ages: 12 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (78):
- Argentina (7):
  - Fundacion Cerebro Y Mente, Mendoza, Mendoza Province
  - Hospital General De Agudos José María Ramos Mejia, Buenos Aires
  - Buenos Aires
  - Centro De Estudio Y Tratamiento De La Epilepsia Y Sueno - Cetes S.A., Córdoba
  - Rosario
  - San José Guaymallén
  - San Miguel de Tucumán
- Australia (5):
  - St Vincent's Hospital Melbourne, Fitzroy
  - Fitzroy
  - Clinical Trials, Epilepsy Research Centre, Melbourne Brain Centre, Heidelberg
  - Royal Melbourne Hospital, Parkville
  - Victoria
- Belgium (5):
  - Uz Antwerpen, Edegem
  - Edegem
  - Uz Gent, Ghent
  - Ghent
  - Ottignies
- Canada (5):
  - Foothills Medical Center, Calgary, Albert
  - London Health Sciences Center, London, Ontario
  - Youthdale Treatment Centers, Toronto, Ontario
  - Calgary
  - London, Ontario
- Chile (5):
  - Puente Alto
  - Hospital Dr. Sótero Del Río, Santiago
  - Santiago
  - Hospital Base Valdivia Servicio De Neurología, Valdivia
  - Valdivia
- Czechia (4):
  - Fakultni Nemocnice U Sv. Anny V Brne, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Ostrava
  - Fakultni Nemocnice V Motole, Prague
- Estonia (5):
  - Laagri
  - West Tallinn Central Hospital, Tallinn
  - Oy Neurodiagnostika Ap, Tallinn
  - Tallinn Children's Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Vantaa, Finland
- Greece, Greece
- Kwai Chung, Hong Kong
- Budapest, Hungary
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Rambam Medical Center, Haifa
  - Haifa
  - Edith Wolfson Medical Center, Holon
  - Netanya
- Italy (2):
  - Azienda Ospedaliera Universitaria Federico Ii, Napoli
  - Napoli
- Latvia (4):
  - Prague
  - Childrens Clinical University Hospital, Riga
  - Riga
  - Outpatient Clinic 'Valmieras Veselibas Centrs', Valmiera
- Lithuania (4):
  - Hospital Of Lithuanian University Of Health Sciences Kaunas Clinics, Kaunas
  - Kaunas
  - Klaipeda University Hospital, Klaipėda
  - Vilnius University Hospital Santariskes Clinics, Vilnius
- Malaysia (2):
  - University Malaya Medical Centre, Kuala Lumpur
  - Petaling Jaya
- Netherlands (3):
  - Haarlem
  - Kempenhaeghe, Heeze
  - Stichting Epilepsie Instellingen Nederland, Hoofddorp
- Poland (2):
  - Akademickie Centrum Kliniczne - Szpital Akademii Medycznej W Gdansku, Gdansk
  - Gdansk
- Spain (8):
  - Albacete
  - Hospital Universitario San Cecilio, Granada
  - Granada
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Madrid
  - Hospital Universitari I Politècnis La Fe Bulevar Sur, Valencia
  - Valencia
- Taiwan (3):
  - Dawan
  - Tainan
  - Taoyuan District
- Thailand (5):
  - King Chulalongkorn Memorial Hospital, Chulalongkorn University, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Bangplee
  - Maharaj Nakorn Chiang Mai, Chiang Mai University, Chiang Mai
  - Srinagarind Hospital, Khonkaen